CLINICAL TRIAL: NCT06376448
Title: An Observational Study Using Novel Questionnaire to Characterize Cough Phenotypes in Patients With Chronic Cough
Status: Recruiting | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: cc-obs-01
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-04

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cough has previously been described by the type of cough you have ie such as wet, dry, and chesty, and also by its features such as how often you are coughing its,intensity, and severity, but never has the varying patterns of cough been studied in any detail and it could be that the pattern of the cough is closely related to patient-perceived intensity, frequency and most importantly severity. Cough is a symptom and like any other symptom (such as pain) the severity of it can only be gauged by the patient experiencing it.

We have created a one-page brand newl questionnaire that shows 4 distinct cough patterns that we believe exist and an empty field designed so that patients can record a pattern of cough they experience which is not already a choice on the questionnaire. The questionnaire also records patients' experience of how frequent, and intense, the cough is, and how it disrupts their lives, on a 1-10 scale (Visual analogue scale), the sum of these scores is collated and this gives us a severity score. The first phase of the project is to determine whether 30 Chronic cough patients understand the questionnaire, and are able to complete it with little direction, and if the cough patterns we identified encompassed all pattern types. second part of the study is to look at how repeatable the questionnaire is when completed over a 6 week period.

DETAILED DESCRIPTION:
STUDY DESIGN This is a single centre observational study.There are two parts to the study. Part 1. Comprises a screening and if suitable the patient will complete the novel questionnaire on one visit.

Part 2. Subjects will be screened, if suitable, patients will be asked to complete the questionnaire and 2-4 weeks later they will be asked to complete the questionnaire once more.

Informed consent and the screening assessment may be conducted either in person at the study site or by telephone, as detailed below.

Informed Consent at Site Potential subjects will be provided with the patient information sheet (PIS) and informed consent form (ICF) at site. A member of the research team will discuss the study with them and take them through the information contained within the PIS and ICF. The subject will be encouraged to ask questions to ensure full understanding. If having read and understood the PIS and ICF the subject wishes to participate, they will sign and date two copies of the ICF, keeping one copy for themselves.

Informed Consent By Telephone

Potential subjects will be sent the PIS and ICF by post or email. Once they have had time to receive and read them, a member of the research team will contact the subject by phone to discuss the study and talk them through the information contained within the PIS and ICF. The subject will be encouraged to ask questions to ensure full understanding. If having read and understood the PIS and ICF the subject gives verbal consent to participate, one of the two following processes will be followed:

* If the full consent discussion has been witnessed at the site, the witness will sign the ICF to confirm that all aspects of the study have been discussed and the subject has freely given verbal informed consent. A copy of the signed ICF will then be sent to the subject.
* If the consent discussion has not been witnessed at the site, the subject will sign and date two copies of the ICF, return one copy to the research team and keep the other copy for themselves.

During screening, eligibility is checked by reference to the selection criteria. If the subject is assessed as eligible for the study, they are assigned a 3-digit subject number. The 3 digit numbers for these patients taking part in part 1, will be prefixed with 1 and those for Part 2, prefixed with a 2.

COUGH PATTERN ASSESSMENTS Part 1. 30 Study participants will be asked to identify their pattern of cough from the patterns identified on the questionnaire, if the patient feels they are unable to identify their pattern then they will be asked to draw a diagram of the pattern and explain the pattern of their cough during the day. This group of patients will be asked to comment on the questionnaire to allow for any improvements. Based on this initial questionnaire completion by this cohort of patients the questionnaire may be updated, especially if new patterns of cough are identified.

Part 2. 30 study participants will be asked to complete the potentially updated questionnaire and then a further copy of the questionnaire will be posted out to these patients for completion 2 to 4 weeks following the first recording on the questionnaire.

Cough frequency/ intensity and disruption Numerical Rating Scale The Cough frequency/ intensity/ and disruption NRS is an 11-point rating scale that patients will be asked to complete.

Each scale is worded as per example below

Now we woud like you to rate how often (frequently) you are coughing , the strength (intensity ) of the cough and overall how disruptive you feel your cough is to your daily life

Please circle most relevant number on scale How often do you cough (Frequency) 0 1 2 3 4 5 6 7 8 9 10 0= no coughing

There are 11 numbered boxes and subjects should select the one that best matches their perception of cough frequency, intensity and disruption to life.

The scores reported on each scale will be summed up to give a total score for severity . This will range from 0-30.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients > 18yrs of age
2. Patients with a current cough of at least 8 weeks duration
3. Patients with a clear chest X-Ray within previous 2 yrs
4. Non- smoker
5. Able to understand and comply with the requirements of the study and sign Informed Consent forms.
6. Good understanding of written and spoken English -

Exclusion Criteria:

1. Recent respiratory tract infection (<4 weeks prior).
2. Current smokers or ex-smokers with <6 months' abstinence prior to Study.
3. Any clinically significant or unstable medical or psychiatric condition that would, in the opinion of the investigator, interfere with the subject's ability to participate in the study safely.
4. Participation in any clinical research study evaluating an investigational drug or therapy within 30 days or within 5 half-lives (whichever is longer) of the investigational drug prior to Study visit. If the subject was in an observational clinical study no washout is required.
5. Subjects who, in the opinion of the Investigator, should not participate in the study for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from those attending the chronic cough clinic or patients that have a history of chronic cough who have previously shown an interest in research.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-10-04 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to characterize and identify the different patterns of cough in chronic cough patients | 1 day
  describe % of various cough patterns recorded and gender differnces and any new patterns

SECONDARY OUTCOMES:
measure of cough severity | 1 day
  To sum up the cough frequency, intensity and disruption to daily life VAS scores to give a measure of cough severity
describe any correlation between severity of cough and cough pattern | 1 day
  To compare cough frequency, intensity and disruption to life with pattern of cough, to determine if any correlation.
reproducibility of questionnnare | 4 weeks
  determine if questionnaire reproducible from repoerting at screening to 4 weeks later

CONTACTS AND LOCATIONS:
Locations (1):
- Redspiratory Medicine, First Floor, Daisy Building, Castle Hill Hospital, Cottingham, East Yorkshiure, United Kingdom